CLINICAL TRIAL: NCT05480085
Title: Screen Free Time With Friends Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Anders Groentved, Professor, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NNF20SH0062965
Record Dates: First submitted 2022-06-21; First posted 2022-07-29 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Screen Media Use; Time With Friends

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School-based extracurricular intervention focusing on screen media use and time spent with friends (Experimental)
  Interventions: Behavioral: School-based extracurricular intervention focusing on screen media use and time spent with friends

INTERVENTIONS:
Behavioral: School-based extracurricular intervention focusing on screen media use and time spent with friends — The intervention includes the following components:
  1. Within each class parents will engage in two meetings combining education and parent-to-parent communication about 1) the children's leisure time activities, and 2) family and class screen time culture. Parents will engage in a short exercise focusing on screen media dilemmas conducted by the teacher in the beginning of 4th grade.
  2. Children will engage in school hour workshops focusing on the class culture related to screen media use and leisure time activities.
  3. Afterschool club personal will engage in mini actions learning program consisting of three workshops aimed to increase participation rate in the afterschool club.
  4. Local stakeholders, e.g., parents, school- and afterschool club personal and others relevant to children's leisure time (e.g., sports clubs) will engage in workshops to adjust the predetermined intervention components (1-3 above) to fit their local context and to develop a local action plan.

SUMMARY:
The Screen Free Time with Friends Feasibility Trial is a study designed to inform development of a definitive trial. The feasibility trial aims to 1) examine the feasibility of an intervention aimed to limit recreational screen media use and promote more time with peers after school and during weekends among 10-11 year old children, 2) examine participant recruitment and retention rates, 3) examine the feasibility of the data collection plan and completeness of the compliance and outcome assessment, and 4) obtain baseline and follow-up data on the planned full trial primary outcome. The Screen Free Time with Friends Feasibility Trial will be conducted as a non-randomized single group feasibility trial including children, their parents and school and afterschool personal from 3rd grade school classes from different schools in the Region of Southern Denmark. The goal is to include a representative sample of children and parents in the participating 3rd grades, and thus there will be no individual level inclusion and exclusion criteria. A process evaluation and outcome measurements will be conducted to evaluate the feasibility and acceptability of the intervention, the data collection plan, and compliance. A baseline- and follow-up assessment will be carried out for some measurements, while others will be collected continuously during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* the distance between the school and the related afterschool club is in walking and cycling distance
* the afterschool club must have potential for improvement (assessed by the municipality)
* the afterschool club personal must have a wish to develop the afterschool club

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | Baseline
  The feasibility of the intervention is evaluated using process evaluation inspired by the RE-AIM framework. Questionnaires to parents and local workshop participants focusing on the intervention and measurements will be used to assess acceptability.
Feasibility of the intervention | After completion of different intervention components
  The feasibility of the intervention is evaluated using process evaluation inspired by the RE-AIM framework. Questionnaires and interviews with parents, local workshop participants, school and afterschool club personal, municipality and research team focusing on the recruitment process, intervention and measurements will be used to assess acceptability.

SECONDARY OUTCOMES:
Participant recruitment and retention rate | Baseline and 6-month follow-up
  Proportion of invited municipalities, schools, afterschool clubs and participants included in the study and proportion of municipalities, schools, afterschool clubs and participants completing the study.
Compliance to leisure time activities measurement | Three times/week for three weeks at baseline and 6-month follow-up
  Proportion of parents answering questions focusing on the child's afterschool club participation and time spent with friends and family during leisure time.
Compliance to objective screen media use measurement | Baseline and 6-month follow-up
  Proportion of children and parents with data on objective measured smartphone use.
Compliance to subjective screen media use measurement | Three times/week for three weeks at baseline and 6-month follow-up
  Proportion of parents answering questions focusing on the child's screen media use during leisure time.
Compliance to objective physical activity measurement | Baseline and 6-month follow-up
  Proportion of children wearing the accelerometer (Axivity AX3) for at least four out of seven measurements days at baseline and follow-up (at least one day must be a weekend day).
Compliance to wellbeing measurement | Baseline and 6-month follow-up
  Proportion of children answering KIDSCREEN-27 questionnaire focusing on wellbeing.
Compliance to a child questionnaire | Baseline and 6-month follow-up
  Proportion of children answering a questionnaire focusing on wellbeing, screen culture in the class and family and children's social relations.
Compliance to a parent questionnaire | Baseline and 6-month follow-up
  Proportion of parents answering the parent questionnaire including questions on background informations, their child's and family's physical activity and screen media habits and children's and parents screen media addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grøntved, PhD, Principal Investigator — Department of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (3):
- Denmark (3):
  - Nyborg municipality, Nyborg
  - Odense municipality, Odense
  - Sorø municipality, Sorø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen SO, Larsen KT, Hoy TV, Hansen ABG, Jago R, Kristensen PL, Toftager M, Grontved A, Gejl AK. Study protocol for the Screen-Free Time with Friends Feasibility Trial. Pilot Feasibility Stud. 2024 Feb 19;10(1):33. doi: 10.1186/s40814-024-01462-y. PMID 38374084